CLINICAL TRIAL: NCT03114722
Title: Citrate 4% Versus Heparinised Saline in Preventing Peripherally Inserted Central Catheter (PICC) Occlusions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016/01420
Record Dates: First submitted 2017-03-20; First posted 2017-04-14 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-03

CONDITIONS: Occlusion
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- heparin 10U/ml (Active Comparator): Heparinised saline (10U/ml) lock in between each catheter use (with standard twice weekly normal saline flushing if catheter not being used)
  Interventions: Drug: Heparinised saline (10U/ml)
- citrate 4% (Experimental): 4% citrate lock in between each catheter use (with standard twice weekly normal saline flushing if catheter not being used)
  Interventions: Drug: Citrate 4%

INTERVENTIONS:
Drug: Citrate 4% — In patients randomised to the citrate arm, the PICC line will be locked with a total of 1.6ml of citrate 4% (0.8ml per lumen in a double-lumen PICC), between each use. Lines will also be flushed with 20ml of normal saline and locked with the locking agent twice a week, if the time elapsed between each use is more than one week. This is part of the standard local protocol. Patients will be followed for up to 6 months or until the catheter is removed, or until the study ends
  Arms: citrate 4%
Drug: Heparinised saline (10U/ml) — In patients randomised to the heparinised saline arm, the PICC line will be locked with 10U/ml heparinised saline between each use. Lines will also be flushed with 20ml of normal saline and locked with the locking agent twice a week, if the time elapsed between each use is more than one week. This is part of the standard local protocol. Patients will be followed for up to 6 months or until the catheter is removed, or until the study ends
  Arms: heparin 10U/ml

SUMMARY:
This study is a prospective, randomized, non-blinded study. 1 group will be assigned the standard arm with use of heparinised saline (10U/ml) lock in between each catheter use. This is consistent with the standard procedure of PICC care in the investigators' centre. The second group will be assigned the intervention with use of 4% citrate lock (Dirinco Citra-Lock 4%) in between each catheter use.

DETAILED DESCRIPTION:
PICC occlusion in patients requiring long-term central line access for chemotherapy is a recurrent issue. Occlusion is usually managed by administration of fibrinolytic agents, and subsequent removal and re-insertion if unsuccessful.

Locally, the current clinical practice is to use heparinised saline at a concentration of 10U/ml as a locking agent in between use of the PICC line to prevent occlusion. Citrate 4% has antithrombotic and antibacterial properties, which makes it potentially superior to heparin as a locking agent. Citrate chelates ionised calcium in blood, inhibiting calcium-dependent clotting pathways. Also, as a chelating agent, it results in inhibition of growth of micro-organisms. Citrate-based anticoagulation is often preferred over heparin because of its safety and rapid systemic clearance. Citrate also is safe for heparin induced thrombocytopenia patients.

The effects of each agent have been compared in renal patients with central lines on haemodialysis. These studies have demonstrated that 4% citrate is at least equivalent (MacRae, 2008) or even superior (Grudzinski, 2007) to heparin 5000U/ml in preventing catheter occlusions, and superior in preventing infection (Weijmer, 2002).

This study is a prospective, randomized, non-blinded study. 1 group will be assigned the standard arm with use of heparinised saline (10U/ml) lock in between each catheter use. This is consistent with the standard procedure of PICC care in the investigators' centre. The second group will be assigned the intervention with use of 4% citrate lock (Dirinco Citra-Lock 4%) in between each catheter use.

Patients will be followed for up to 6 months or until the catheter is removed, or until the study ends. A standardised data tracking form will be used to assess baseline characteristics as well as number of times urokinase was used. Nursing documentation regarding each PICC flushing (standard documentation as per hospital protocol) will be evaluated for number of discrete attempts made to troubleshoot lines without use of urokinase. Positive blood culture results will be recorded for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal to 21 years.
* Histologic or cytologic diagnosis of haematological or oncological malignancy
* Signed informed consent from patient or legal representative
* Patients on antiplatelet therapy may be recruited to the study

Exclusion Criteria:

* Pregnancy.
* Anticoagulation - warfarin or heparin or novel oral anticoagulants
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-07-31 (Estimated); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of catheter occlusion | From post insertion to 6 months or until the catheter is removed, whichever is earlier.
  Compare the rates of catheter occlusion in patients who receive citrate 4% as a locking agent, versus those who receive heparinised saline (10U/ml).

SECONDARY OUTCOMES:
Line troubleshooting | From post insertion to 6 months or until the catheter is removed, whichever is earlier.
  to compare the time to requiring troubleshooting of the line but not amounting to urokinase use
Catheter associated bacteraemia | From post insertion to 6 months or until the catheter is removed, whichever is earlier.
  to compare the time to development of catheter associated bacteraemia
Bleeding complications | From post insertion to 6 months or until the catheter is removed, whichever is earlier.
  to compare the time to development of bleeding complications, either local or systemic.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Nationa University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macrae JM, Dojcinovic I, Djurdjev O, Jung B, Shalansky S, Levin A, Kiaii M. Citrate 4% versus heparin and the reduction of thrombosis study (CHARTS). Clin J Am Soc Nephrol. 2008 Mar;3(2):369-74. doi: 10.2215/CJN.01760407. PMID 18308996
- [Background] Grudzinski L, Quinan P, Kwok S, Pierratos A. Sodium citrate 4% locking solution for central venous dialysis catheters--an effective, more cost-efficient alternative to heparin. Nephrol Dial Transplant. 2007 Feb;22(2):471-6. doi: 10.1093/ndt/gfl606. Epub 2006 Oct 25. PMID 17065193
- [Background] Weijmer MC, Debets-Ossenkopp YJ, Van De Vondervoort FJ, ter Wee PM. Superior antimicrobial activity of trisodium citrate over heparin for catheter locking. Nephrol Dial Transplant. 2002 Dec;17(12):2189-95. doi: 10.1093/ndt/17.12.2189. PMID 12454232
- [Background] Strauss RG. Mechanisms of adverse effects during hemapheresis. J Clin Apher. 1996;11(3):160-4. doi: 10.1002/(SICI)1098-1101(1996)11:33.0.CO;2-9. PMID 8915821